CLINICAL TRIAL: NCT03814876
Title: Effect of a Manualized Family Intervention Following Brain Injury or Spinal Cord Injury
Brief Title: Family Intervention Following Traumatic Injury
Acronym: FITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Danish Victims Fund (Other Government); The Association of Eastern Founders (Other)
Responsible Party: Principal Investigator, Anne Norup, Principle investigator, neuropsychologist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018_0004
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acquired Brain Injury; Spinal Cord Injuries
MeSH Terms: conditions — Brain Injuries; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCI intervention (Experimental): Spinal cord injury intervention group
  Interventions: Behavioral: FITS
- SCI control (Active Comparator): Spinal cord injury control
  Interventions: Behavioral: Group session psycho-education
- TBI intervention (Experimental): Traumatic brain injury intervention group
  Interventions: Behavioral: FITS
- TBI control (Active Comparator): Traumatic brain injury control group
  Interventions: Behavioral: Group session psycho-education

INTERVENTIONS:
Behavioral: Group session psycho-education — Active comparator - control group
  Arms: SCI control; TBI control
Behavioral: FITS — Manualized family intervention
  Arms: SCI intervention; TBI intervention

SUMMARY:
The purpose of this study is to investigate the effectiveness of a manualized intervention (FITS) to families living with brain injury or spinal cord injury. The intervention will be provided by a trained neuropsychologist and consists of 8 structured sessions of 90 minutes duration. The intervention group will be compared to a control group receiving treatment as usual, one psycho-educational group session of a 2 hour duration.

ELIGIBILITY:
Inclusion Criteria:

* Acquired brain injury or spinal cord injury
* Talk and read Danish
* Minimum 6 months to 2 years since discharge
* Family members must be actively involved in the patient's rehabilitation

Exclusion Criteria:

* Severe aphasia
* Families, where other family members require a substantial amount of care
* Prior psychiatric or neurological disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Disease specific quality of life | Change from day 0 to week 8, follow up at six months
  Measured by Qolibri for patients with traumatic brain injury. The QOLIBRI consists of six novel items that assess overall satisfaction with facets of life relevant to people with TBI. Areas covered by the questionnaire include physical condition, cognition, emotions, function in daily life, personal and social life, and current situation and future prospects. Responses to each item are scored 1 ('Not at all') to 5 ('Very'), and the sum of all items was converted arithmetically to a percentage scale, with 0 representing the lowest possible HRQoL on the questionnaire and 100 the best possible HRQoL.
Generic quality of life | Change from day 0 to week 8, follow up at six months
  Short Form-36 (SF-36) completed by all participants. SF-36, a measure of self-reported HRQoL. The questionnaire comprises 36 items addressing eight dimensions of health: vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health. The original summative scoring algorithm will be used, and raw scores will be converted into standard SF-36 scores ranging from 0-100 by calculating the product 100∗(actual sum score / highest possible score), with higher scores indicating better health. The scores will be evaluated according to Danish norms provided by Bjorner, Damsga°rd, Watt, and Bech (1997). This normative study showed high Cronbach's alpha coefficients on all the sub-scales ranging from .75-.85 (Bjorner et al., 1997).
Disease specific quality of life | Change from day 0 to week 8, follow up at six months
  QoL basic data elements for spinal cord injury for patients with spinal cord injury. The QoL Basic Data Set consists of three items on satisfaction with life as a whole, satisfaction with physical health and satisfaction with psychological health during the past 4 weeks. Each item is answered on a 0-10 numerical rating scale with markers 'complete dissatisfaction' and 'complete satisfaction'.
Caregiver burden | Change from day 0 to week 8, follow up at six months
  Caregiver burden questionnaire. The burden of the caregivers will be assessed using the 22-item scale Caregiver Burden (CB). The scale consists of five sub-scales: General Strain, Isolation, Disappointment, Emotional Involvement and Environment. A Total Burden index is given by calculating the mean of all 22 items. Each of the 22-items is scored 1-4 (Not at all, Seldom, Sometimes, Often) and the items cover aspects such as caregiver health, psychological well-being, relationship, social network, physical workload and environmental aspects.
Self-perceived burden | Change from day 0 to week 8, follow up at six months
  Burden perceived by the patient (SPB). The patients' SPB was measured with the Danish version of Self-Perceived Burden Scale (SPBS), which contains 10 items and scores range from 0-50. The 10 items were selected based on one single, general burden factor (Cousineau et al. 2003). Higher scores indicate high SPB. To estimate how severe self-perceived burden did patients feel, SPBS scores can be categorised into four stages: none to little (≤ 19), mild to moderate (20-29),moderate to severe (30-39) and severe (≥40).

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Langer Soendergaard, MSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Stevens LF, Lehan T, Duran MAS, Plaza SLO, Arango-Lasprilla JC. Pilot Study of a Newly Developed Intervention for Families Facing Serious Injury. Top Spinal Cord Inj Rehabil. 2016 Winter;22(1):49-59. doi: 10.1310/sci2201-49. PMID 29398893
- [Derived] Soendergaard PL, Wolffbrandt MM, Biering-Sorensen F, Nordin M, Schow T, Arango-Lasprilla JC, Norup A. A manual-based family intervention for families living with the consequences of traumatic injury to the brain or spinal cord: a study protocol of a randomized controlled trial. Trials. 2019 Nov 27;20(1):646. doi: 10.1186/s13063-019-3794-5. PMID 31775831